CLINICAL TRIAL: NCT01091558
Title: Immunomodulary Effects of Arginine Supplementation in Colitis and Colon Cancer
Brief Title: Study of Effects of L-Arginine in Colitis and Colon Cancer
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Keith Wilson, Professor of Medicine, Vanderbilt University Medical Center
Other Study IDs: 090943; 3R01AT004821-02S1 (NIH)
Record Dates: First submitted 2010-03-18; First posted 2010-03-24 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Ulcerative Colitis; Colon Cancer
Keywords: ulcerative colitis; colon cancer; endoscopy; screening
MeSH Terms: conditions — Colitis, Ulcerative; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, urine and tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Colonoscopy: Healthy volunteer who is having a screening colonoscopy
- Ulcerative Colitis: Patients with confirmed ulcerative colitis who are scheduled for endoscopy for medical reasons.

SUMMARY:
The purpose of this study is to look at the importance of L-Arginine in the digestive tract. L-Arginine is an amino acid and is important in making proteins within the cell.

The evaluation of colon tissue, blood, urine, diet, health history, and symptoms will help us learn more about L-Arginine and ulcerative colitis. The investigators believe these studies will provide new insights into the treatment for Inflammatory Bowel Disease (ulcerative colitis) and nutritional needs. The investigators plan to enroll 200 participants in this study over the next two years.

DETAILED DESCRIPTION:
Amino acids are being measured in colon tissues and in serum by high performance liquid chromotography (HPLC). Cytokines and chemokines are being measured in colon tissues and in serum by Luminex assay. Cytokines and chemokines are also being measured in colon tissues by real-time polymerase chain reaction (PCR) analysis of mRNA expression.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Colonoscopy for one of the following: clinical indications, disease assessment, or surveillance for dysplasia (as in ulcerative colitis)
* Screening for cancer

Exclusion Criteria:

* refusal to participate
* age less than 18 years at time of colonoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any patient scheduled to have a colonoscopy as part of medical care for either ulcerative colitis or as a routine screening colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
L-Arginine (L-Arg) availability in ulcerative colitis (UC) patients and normal control subjects, and correlate with disease activity | 24 months

SECONDARY OUTCOMES:
L-Arg intake in the diet of UC patients and control subjects | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Keith Wilson, MD, AGAF, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Hospital, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gobert AP, Latour YL, Asim M, Barry DP, Allaman MM, Finley JL, Smith TM, McNamara KM, Singh K, Sierra JC, Delgado AG, Luis PB, Schneider C, Washington MK, Piazuelo MB, Zhao S, Coburn LA, Wilson KT. Protective Role of Spermidine in Colitis and Colon Carcinogenesis. Gastroenterology. 2022 Mar;162(3):813-827.e8. doi: 10.1053/j.gastro.2021.11.005. Epub 2021 Nov 10. PMID 34767785